CLINICAL TRIAL: NCT00006384
Title: Phase II Trial of SU5416 and Interferon Alfa 2B in Unresectable or Metastatic Renal Cell Carcinoma
Brief Title: SU5416 and Interferon Alfa-2b in Treating Patients With Unresectable or Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 00041; U01CA062505 (NIH); P30CA033572 (NIH); CHNMC-PHII-23; NCI-T99-0085; CDR0000068262 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2000-10-04; First posted 2003-12-24 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Interferon-alpha; Semaxinib

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: semaxanib

SUMMARY:
RATIONALE: SU5416 may stop the growth of kidney cancer by stopping blood flow to the tumor. Interferon alfa-2b may interfere with the growth of the cancer cells. Combining interferon alfa-2b with SU5416 may be an effective treatment for kidney cancer.

PURPOSE: Phase II trial to study the effectiveness of combining SU5416 and interferon alfa-2b in treating patients who have unresectable or metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy and toxicity of SU5416 combined with interferon alfa-2b in patients with unresectable or metastatic renal cell carcinoma.

OUTLINE: This is a multicenter study. Patients receive SU5416 IV over 30-60 minutes twice weekly and interferon alfa-2b subcutaneously every 12 hours daily. Treatment continues every 6 weeks for a minimum of 2 courses. Patients who achieve partial response or stable disease after completion of course 2 receive additional courses in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response may receive additional courses, at the discretion of the protocol investigator, in the absence of disease progression or unacceptable toxicity. Patients with disease progression are allowed to stay on the study until any measurable lesion increases to over 100% of baseline measurement. Patients are followed for survival.

PROJECTED ACCRUAL: A total of 20-31 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed unresectable or metastatic renal cell carcinoma Measurable or evaluable disease Prior nephrectomy allowed if documented disease progression prior to study No known brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: WBC at least 3,500/mm3 Absolute granulocyte count at least 1,500/mm3 Platelet count at least lower limit of normal Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT no greater than 2 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No uncompensated coronary artery disease by ECG or physical examination No myocardial infarction or severe/unstable angina within the past 6 months No severe peripheral vascular disease associated with diabetes mellitus No deep venous or arterial thrombosis within the past 3 months Pulmonary: No pulmonary embolism within the past 3 months Other: No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix Not pregnant or nursing Fertile patients must use effective contraception No documented hypersensitivity to any excipients (Cremophor EL, ethanol, or polyethylene glycol) of SU5416

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 8 weeks since prior interleukin-2 and recovered No other prior biologic therapy Chemotherapy: At least 4 weeks since prior chemotherapy and recovered No more than 1 prior chemotherapy regimen Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy No concurrent radiotherapy to measurable lesions Surgery: See Disease Characteristics More than 3 weeks since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-11; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Primo N. Lara, MD, Study Chair — University of California, Davis
Locations (3):
- United States (3):
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California

REFERENCES:
- [Result] Lara PN Jr, Quinn DI, Margolin K, Meyers FJ, Longmate J, Frankel P, Mack PC, Turrell C, Valk P, Rao J, Buckley P, Wun T, Gosselin R, Galvin I, Gumerlock PH, Lenz HJ, Doroshow JH, Gandara DR; California Cancer Consortium. SU5416 plus interferon alpha in advanced renal cell carcinoma: a phase II California Cancer Consortium Study with biological and imaging correlates of angiogenesis inhibition. Clin Cancer Res. 2003 Oct 15;9(13):4772-81. PMID 14581348